CLINICAL TRIAL: NCT06653894
Title: Evaluation of the Postoperative Analgesic Efficacy of Pericapsular Nerve Group (PENG) Block and Quadratus Lumborum Block (QLB) in Hip Surgeries
Brief Title: Postoperative Analgesic Efficacy of PENG and QLB Blocks in Hip Surgeries
Acronym: PENG vs QLB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, SERPİL ŞEHİRLİOĞLU, Anesthesiology and Reanimation Specialist, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREH-PENG
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-05

CONDITIONS: Hip Surgery; Postoperative Analgesia
Keywords: PENG; QLB; Postoperative Analgesia; Hip Surgery
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QLB Group (Active Comparator): In the QLB (Quadratus Lumborum Block) group, patients will be placed in the lateral decubitus position, and the block will be performed using ultrasound guidance
  Interventions: Procedure: anterior quadratus lumborum block
- PENG Block Group (Active Comparator): In the PENG (Pericapsular Nerve Group) block group, patients will be positioned supine, and the block will be performed under ultrasound guidance.
  Interventions: Procedure: PENG block with 0.25% bupivacaine.

INTERVENTIONS:
Procedure: PENG block with 0.25% bupivacaine. — In the PENG group, patients were placed in the supine position. A convex ultrasound probe was positioned under sterile conditions on the operated side, aligned with the iliac bone below the anterior superior iliac spine (ASIS). The anterior inferior iliac spine (AIIS), iliopubic eminence (IPE), iliopsoas muscle, and its tendon were identified. Using an in-plane technique, a 22G 100-mm peripheral block needle was advanced toward the IPE, targeting the space between the iliopsoas muscle tendon and the IPE. Proper placement was confirmed via hydrodissection. Subsequently, 20 mL of 0.25% bupivacaine was administered slowly, with aspiration performed every 5 mL to avoid intravascular injection. The correct spread of the local anesthetic was verified via ultrasound, confirming elevation of the iliopsoas tendon.
  Arms: PENG Block Group
Procedure: anterior quadratus lumborum block — The quadratus lumborum and psoas major muscles, along with the transverse process of the L4 vertebra, were visualized in the midaxillary line using an in-plane technique. A 22G, 100-mm peripheral block needle (Stimuplex® Ultra; B. Braun Melsungen AG, Melsungen, Germany) was advanced into the subfascial plane between the quadratus lumborum and psoas major muscles, and 1-2 mL of 0.9% saline was injected to confirm correct placement via hydrodissection.
  Following this, 20 mL of 0.25% bupivacaine (Buvasin® 0.5%, VEM, Tekirdağ, Turkey) was injected incrementally, with aspiration performed every 5 mL. Proper spread of the local anesthetic was confirmed by ultrasound visualization of a hypoechoic distribution between the fascial planes.
  Arms: QLB Group

SUMMARY:
This prospective, randomized, single-blinded study compares the postoperative analgesic efficacy of the Pericapsular Nerve Group (PENG) block and Quadratus Lumborum Block (QLB) in hip surgeries under spinal anesthesia. the study focuses on time to first rescue analgesia and total analgesic consumption within the first 48 hours postoperatively in patients over 40 years undergoing elective hip surgery. Ninety patients will be randomized into two groups (PENG or QLB) using a sealed envelope method. The study will assess pain scores, opioid consumption, and side effects, hypothesizing that both blocks provide effective analgesia but seek to identify which offers superior efficacy. Statistical analysis will be performed with SPSS, aiming to contribute valuable insights into analgesic techniques for hip surgeries.

DETAILED DESCRIPTION:
This is a prospective, randomized single-blinded study comparing the postoperative analgesic efficacy of Pericapsular Nerve Group (PENG) block and Quadratus Lumborum Block (QLB) in hip surgeries performed under spinal anesthesia. The study aims to evaluate key outcomes such as the time to first rescue analgesia and total analgesic consumption within the first 48 hours postoperatively. The primary population includes patients over 40 years undergoing elective hip surgery with specific inclusion and exclusion criteria. ninety patients will be divided into two groups, receiving either QLB or PENG block, using a sealed envelope randomization method.

PENG block targets specific nerves to provide analgesia without motor block, preserving motor function. QLB involves injecting a local anesthetic into the fascia near the quadratus lumborum muscle to block thoracoabdominal nerves and provide broad analgesia. Data on pain scores (NRS), opioid consumption, and side effects will be collected at different time points.

The study hypothesizes that both blocks can provide effective postoperative analgesia, with potential benefits such as reduced opioid consumption , but aims to determine which block is superior in efficacy.

The primary aim of this study was to compare the effect of an anterior QLB and PENG block on total opioid analgesic consumption within the first 48 hours postoperatively. The secondary aims were to compare the resting and dynamic NRS scores at 2, 12, 24 and 48 hours postoperatively, the time to first rescue analgesia, and side effects such as nausea, vomiting and quadriceps weakness.

Statistical analysis will be conducted using SPSS, and findings will contribute to the literature on analgesia techniques for hip surgeries.

ELIGIBILITY:
Inclusion Criteria:

* "Patients aged over 40 years who are scheduled to undergo hip surgery under spinal anesthesia and classified as ASA 1-3 will be included in the study."

Exclusion Criteria:

* Patients who refuse the procedure.
* Patients who will receive general anesthesia or peripheral nerve blocks such as a combination of femoral and sciatic nerve blocks.
* A history of allergy to local anesthetic agents.
* Patients with a diagnosis of neurocognitive disorders such as dementia or Alzheimer's disease under active neurological follow-up.
* Patients with multiple trauma.
* Patients with severe hearing or vision impairments.
* Patients with a local infection at the site of the block application.
* Patients with a Body Mass Index (BMI) > 35.
* Patients with a history of severe neurological, cardiovascular, renal, or hepatic disease will be excluded from the study.
* Patients who, during the postoperative period, required intensive care unit (ICU) admission for more than one day due to hemodynamic monitoring or sedation, as well as those who developed complications during postoperative follow-up-such as re-operation, postoperative hemorrhage, or the need for advanced cardiopulmonary support-were excluded from the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Total Opioid Consumption | 48 hour
  Total Opioid Consumption

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) Scores | 48 hour
  Assessed at various time points to quantify pain intensity at rest and during movement. The Numerical Rating Scale (NRS) is a pain assessment tool where patients rate their pain from 0 (no pain) to 10 (worst pain).
Time to First Rescue Analgesic | 48 hours
  Duration from the end of surgery to the first request for analgesic medication.
Adverse Events | 48 hour
  Monitoring for complications or side effects related to the nerve blocks

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stuart Green M, Ryan Hoffman C, Iqbal U, Olabisi Ives O, Hurd B. Transmuscular Quadratus Lumborum Block Reduces Length of Stay in Patients Receiving Total Hip Arthroplasty. Anesth Pain Med. 2018 Nov 20;8(6):e80233. doi: 10.5812/aapm.80233. eCollection 2018 Dec. PMID 30719411
- [Background] Farag A, Hendi NI, Diab RA. Does pericapsular nerve group block have limited analgesia at the initial post-operative period? Systematic review and meta-analysis. J Anesth. 2023 Feb;37(1):138-153. doi: 10.1007/s00540-022-03129-5. Epub 2022 Nov 7. PMID 36342537
- [Background] Zheng J, Pan D, Zheng B, Ruan X. Preoperative pericapsular nerve group (PENG) block for total hip arthroplasty: a randomized, placebo-controlled trial. Reg Anesth Pain Med. 2022 Mar;47(3):155-160. doi: 10.1136/rapm-2021-103228. Epub 2021 Dec 6. PMID 34873023